CLINICAL TRIAL: NCT05479305
Title: Evaluation of the Valiant Captivia Physician Fenestrated Stent Graft System in Aortic Arch and Descending Thoracic Aorta Pathologies
Acronym: EVERGREEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ceric Sàrl (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVERGREEN
Record Dates: First submitted 2022-07-25; First posted 2022-07-29 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Penetrating Ulcer of Aorta; Aneurysm Aortic; Type B Aortic Dissection; Residual Dissection After Type A Repair
Keywords: aortic arch; descending thoracic aorta; valiant captivia stent graft
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention/Treatment (Experimental): The Valiant Captivia physician fenestrated stent graft for the treatment of aneurysms/penetrating ulcers, Type B aortic dissections or residual dissection after Type A repair, of the aortic arch and the descending thoracic aorta which are candidates for revascularisation of all three supra-aortic vessels (BT, LCCA, LSA)
  Interventions: Device: The Valiant Captivia Stent Graft

INTERVENTIONS:
Device: The Valiant Captivia Stent Graft — Aortic arch/Descending aorta Repair

SUMMARY:
The study objectives are to assess safety and effectiveness, measured acutely and at the 30-day visit after implantation of the Valiant Captivia physician fenestrated Stent Graft.

Clinical utility measures throughout the procedure and until discharge will be assessed

DETAILED DESCRIPTION:
Prospective, single-arm, non-randomised, multicenter, investigator initiated clinical study evaluating subjects implanted with The Valiant Captivia physician fenestrated stent graft for the treatment of aneurysms/penetrating ulcers, Type B aortic dissections or residual dissection after Type A repair, of the aortic arch and the descending thoracic aorta which are candidates for revascularisation of all three supra-aortic vessels (BT (brachiocephalic trunk) , LCCA (left Common Carotid artery), LSA (Left Subclavian Artery)

ELIGIBILITY:
Inclusion Criteria:

TAA/PAU (Thoracic Aortic Aneurysms and Penetrating Ulcers):

1. Subject is at least 18 years of age.
2. Subject understands and has signed an Informed Consent approved by the Sponsor for this study.
3. Subject must be considered a candidate for revascularisation of BT, LCCA and LSA.
4. Subject must be able to tolerate surgical revascularisation of BT, LCCA and LSA.
5. Subject has a TAA/PAU which is:

   * a fusiform aneurysm with a diameter of ≥ 5.5 cm OR is > 2 times the diameter of the non-aneurysmal thoracic aorta; AND/OR
   * a saccular aneurysm or PAU (ulcer defined as ≥ 10 mm in depth and 20 mm in diameter, or symptomatic)
6. Subject has a healthy, non-diseased aortic proximal seal zone of at least 20 mm
7. Subject has no thrombus in the proximal neck
8. Subject has a non-diseased aortic diameter between 25 mm and 42 mm and max diameter of the ascending aorta is ≤ 40 mm
9. Subject has a non-diseased LSA which is eligible for stent-grafting
10. Subject has sufficient landing zone within the LSA to accommodate the stent-graft without occlusion of any significant vessels
11. Brachial, iliac or femoral artery access vessel morphology (diameter, calcification, tortuosity) that is compatible with vascular access techniques, the device, or accessories.
12. Symptomatic patient who needs semi urgent repair; aptient is at high surgical risk and cannot wait for 6-8 weeks for a custom-made stent graft
13. Subject is affiliated with the social security system

Inclusion criteria:

TBAD(Type B Dissections) and Residual dissection after Type A repair:

1. Subject is at least 18 years of age.
2. Subject understands and has signed an Informed Consent approved by the Sponsor for this study.
3. a) Subject has a degenerative aortic arch aneurysm which will require coverage of the LSA and extension of the proximal seal zone to zone 0 And/or b) Subject has a complicated TBAD (acute, subacute or chronic) which will require coverage of the LSA and extension of the proximal seal zone to zone 0 And/or c) Subject has a complicated residual dissection after replacement of the ascending aorta for type A aortic dissection which will require coverage of the LSA and extension of the proximal seal zone to zone 0
4. Subject has a healthy, non-diseased (without thrombus) aortic proximal seal zone of at least 20 mm
5. Subject has a healthy, non-diseased (without thrombus) aortic distal seal zone of at least 20 mm
6. Subject has a maximum diameter of the distal ascending aorta just above the BT of 40 mm
7. Subject has a non-diseased aortic diameter between 28 mm to 42 mm and the ascending aorta ≤ 40 m
8. Subject has a no atheromatous lesions int the arch and the BT, LCCA and LSA
9. Brachial, iliac or femoral artery access vessel morphology (diameter, calcification, tortuosity) that is compatible with vascular access techniques, the device, or accessories
10. Symptomatic patient who needs semi urgent repair; aptient is at high surgical risk and cannot wait for 6-8 weeks for a custom-made stent graft
11. Subject is affiliated with the social security system

Exclusion Criteria:

(Thoracic Aortic Aneurysms and Penetrating Ulcers, TAA/PAU):

1. Subject has an aneurysmal, tortuous, or atherosclerotic LSA.
2. Subject has an aneurysmal, tortuous, or atherosclerotic LCCA.
3. Subject has an aneurysmal, tortuous, or atherosclerotic BT.
4. Subject has an ascending aorta diameter > 40 mm
5. Subject has thrombus in the proximal neck
6. Subject has an emergent need of treatment of the aortic pathology
7. Subject has prohibitive calcification, occlusive disease, or tortuosity of intended sealing sites
8. Subject has circumferential calcification in the common femoral or external iliac artery or in the common iliac artery with an intraluminal diameter (ID) less than 9 mm at any point proximal to or at the access vessel site unless a surgical adjunctive procedure is planned.
9. Subject has an aortic atheroma classified as grade IV or grade V.
10. Subject has had previous endovascular repair of the ascending
11. Subject has significant and/or circumferential aortic mural thrombus at either the proximal or distal attachment sites that would compromise sealing of the device.
12. Subject is pregnant
13. Subject has a known allergy or intolerance to the device components.
14. Subject is in acute renal failure
15. Subject has a body habitus which prevents adequate visualisation of the aorta.
16. Subject has coronary artery disease with unstable angina and who has not received treatment.
17. Subject has a connective tissue disease (e.g. Marfan's syndrome, medial degeneration).
18. Subject has active systemic infection and/or a mycotic aneurysm.
19. Subject is currently participating in an investigational drug or device clinical trial that would interfere with the observations of this study.
20. Subject has other medical, social, or psychological problems that, in the opinion of the investigator, will interfere with treatment and follow-up procedures.
21. Subject has a life expectancy of less than 2 years year.
22. Subject requires treatment of an infrarenal aneurysm at the time of the implantation.
23. Subject has had previous surgical or endovascular treatment of an infra-renal aortic aneurysm <30 days of implantation of investigational device.
24. Subject has a history of bleeding diathesis, coagulopathy, or refuses blood transfusion.
25. Subject has had a cerebral vascular accident (CVA) within 3 months.
26. Subject has had a myocardial infarction (MI) within 3 months.
27. Subject has a known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment

Exclusion criteria:

(Type B Dissections, TBAD and residual dissection after Type A repair):

1. Subject has an aneurysmal, tortuous, or atherosclerotic LCCA.
2. Subject has an aneurysmal, tortuous, or atherosclerotic LSA.
3. Subject has an aneurysmal, tortuous, or atherosclerotic BT.
4. Subject has a dissected BT and or LCCA
5. Subject has prohibitive calcification, occlusive disease, or tortuosity of intended sealing sites.
6. Subject has circumferential calcification in the common femoral artery, external iliac artery or in the common iliac artery with an intraluminal diameter (ID) less than 9 mm at any point proximal to or at the access vessel site unless a surgical adjunctive procedure is planned.
7. Subject has an aortic atheroma classified as grade IV or grade V.
8. Subject has had previous endovascular repair of the ascending, arch
9. Subject has significant and/or circumferential aortic mural thrombus at either the proximal or distal sealing sites that would compromise seal of the device
10. Subject is pregnant
11. Subject has a known allergy or intolerance to the device components
12. Subject is in acute renal failure
13. Subject has a body habitus which prevents adequate visualisation of the aorta.
14. Subject has coronary artery disease with unstable angina and who has not received treatment.
15. Subject has a connective tissue disease (e.g. Marfan's syndrome, medial degeneration).
16. Subject has active systemic infection and/or a mycotic aneurysm.
17. Subject is currently participating in an investigational drug or device clinical trial that would interfere with the observationsof this study
18. Subject has other medical, social, or psychological problems that, in the opinion of the investigator, will interfere with treatment and follow-up procedures.
19. Subject has a life expectancy of less than 2 years.
20. Subject requires treatment of an infrarenal aneurysm at the time of the implantation.
21. Subject has had previous surgical or endovascular treatment of an infra-renal aortic aneurysm <30 days of implantation of investigational device.
22. Subject has a history of bleeding diathesis, coagulopathy, or refuses blood transfusion.
23. Subject has had a cerebral vascular accident (CVA) within 3 months.
24. Subject has had a myocardial infarction (MI) within 3 months.
25. Subject has a known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoints: | 30 days
  Within one month (Day 0 - Day 30) from the index procedure, composite endpoint consisting of:
  * Aorta-Related Mortality
  * Stroke/TIA (Transient Ischemic Attack)
  * Paraplegia/paraparesis
  * Left Arm/Hand Ischemia
Primary Effectiveness Endpoints: | 30 days
  The primary effectiveness endpoint is treatment success (defined below) and will be captured within the initial reporting period of 1 month from the index procedure.
  Treatment success defined as technical success comprising the following:
  * the successful delivery and deployment of the stent graft (The Valiant Captivia physician fenestrated Stent Graft) at the planned location
  * no unintentional coverage of supra-aortic vessels, assessed intra-operatively,
  * the removal of the delivery system
  * successful exclusion of the aortic lesion while maintaining patency of the LSA stent-graft as well as LCCA and BT at the 30-day visit

SECONDARY OUTCOMES:
Intra/periprocedural through Discharge Clinical Utility Measures 1 | 0 to 30 days
  Mean duration (min) of the procedure.
Intra/periprocedural through Discharge Clinical Utility Measures 2 | 0 to 30 days
  • Mean time (min) to implant
Intra/periprocedural through Discharge Clinical Utility Measures 3 | 0 to 30 days
  Proportion of subjects who underwent general anaesthesia.
Intra/periprocedural through Discharge Clinical Utility Measures 4 | 0 to 30 days
  Mean volume (cc) of estimated blood loss.
Intra/periprocedural through Discharge Clinical Utility Measures 5 | 0 to 30 days
  Proportion of subjects requiring blood transfusion
Intra/periprocedural through Discharge Clinical Utility Measures 6 | 0 to 30 days
  Mean length of time (days) of overall hospital stays
Intra/periprocedural through Discharge Clinical Utility Measures 7 | 0 to 30 days
  Mean length of time (hours) in the intensive care unit.
Major adverse event | Up to 3 years
  All-Cause Mortality
  * Myocardial Infarction
  * Paraplegia/Paraparesis
  * Renal Failure
  * Stroke/TIA
  * Left Arm/Hand Ischemia
Secondary endovascular procedures | Up to 3 years
  repeating procedures
Secondary endovascular procedures for primary device failures | Up to 3 years
  (including Type I/III endoleaks, aneurysm expansion, aneurysm/aortic rupture, and supra-aortic vessels including LSA stent-graft occlusion)
Other | Up to 3 years
  * Rupture
  * Endoleaks
  * Maximum aneurysm diameter changes from baseline*
  * Exclusion of aneurysm
  * Exclusion of penetrating aortic ulcer (PAU)
  * Stent graft patency
  * Stent graft integrity
  * Conversion to surgical repair
  * Surgical revascularisation of the LSA, LCCA, BT
  * Paraparesis
  * Adverse events including serious adverse events and device, procedure, and/or disease-related adverse events
For TBAD, these additional observations will be evaluated | 0 to 30 days
  Coverage of primary entry tear (exclusion of false lumen)
  * Extension of dissection (proximally or distally) with or without complications
  * Continuing or new false lumen (FL) perfusion
  * Aortic remodeling post-procedure

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CH de Brest, Brest
  - Hôpital Louis Pradel, Bron
  - CHU de Montpellier, Montpellier
  - CH d'Orléans, Orléans

IPD SHARING:
Plan to Share IPD: No